CLINICAL TRIAL: NCT05555147
Title: The Effect of Bilateral Infraorbital and Infratrochlear Nerve Block on Perioperative Analgesia After Endoscopic Binostril Transnasal Transsphenoidal Resection of Pituitary: a Prospective, Randomized Study
Brief Title: The Effect of Bilateral Infraorbital and Infratrochlear Nerve Block on Perioperative Period of Hypophysectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Feng Gao, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TJ2012S152
Record Dates: First submitted 2022-03-01; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Pain; Nerve Block
MeSH Terms: conditions — Pain | interventions — Nerve Block; Ropivacaine

STUDY DESIGN:
Intervention Model Description: Thirty minutes prior to surgery the patients received bilateral infraorbital and infratrochlear nerve block. The patient's head was positioned on a central line in the supine position. A 25 gauge needle was inserted laterally to the ipsilateral nostril after palpating the infraorbital ridge to locate the infraorbital foramen. The index finger of the non-dominant hand was positioned above the infraorbital foramen, and the needle was advanced until it was felt beneath the finger . 2 mL of the study solution was slowly injected after negative aspiration of blood was confirmed. Inserting the needle 1 cm above the inner canthus, targeting the junction of the orbit and the nasal bone, performed Infratrochlear nerve block. After negative aspiration of blood, 1 mL of the study solution was injected. Contralateral nerve block was performed in the same manner.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients were randomly assigned to one of two groups by a single nurse, who was not involved in the anesthetic management of the patient, while using a computer-generated randomization sequence with random block sizes of two and four. The same nurse prepared syringes containing the nerve block solution. Syringes for the block group (Block group) were filled with 6 mL of 0.5% ropivacaine. The patient, surgeon,and investigator were all blinded to the study and the adequacy of the block.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve Block Group (Experimental): Thirty minutes prior to surgery the patients received bilateral infraorbital and infratrochlear nerve block. Infraorbital nerve block was performed while using an extraoral approach. A 25 gauge needle was inserted laterally to the ipsilateral nostril after palpating the infraorbital ridge to locate the infraorbital foramen. The index finger of the non-dominant hand was positioned above the infraorbital foramen, and the needle was advanced until it was felt beneath the finger. 2 mL of the 0.5% ropivacaine slowly injected after negative aspiration of blood was confirmed. Inserting the needle 1 cm above the inner canthus, targeting the junction of the orbit and the nasal bone, performed Infratrochlear nerve block. After negative aspiration of blood, 1 mL of the 0.5% ropivacaine was injected. Contralateral nerve block was performed in the same manner.
  Interventions: Drug: nerve block with 0.5% ropivacaine
- Control Group (Sham Comparator): Patients receiving general anesthesia without Infraorbital and Infratrochlear nerve block.
  Interventions: Other: without any nerve block

INTERVENTIONS:
Drug: nerve block with 0.5% ropivacaine — After general anesthesia, the patients will receive bilateral infraorbital and infratrochlear nerve block 30 minutes prior to surgery. Infraorbital nerve block is performed while using an extraoral approach. A 25-gauge needle was inserted laterally to the ipsilateral nostril after palpating the infraorbital ridge to locate the infraorbital foramen. The index finger of the non-dominant hand was positioned above the infraorbital foramen, and the needle was advanced until it was felt beneath the finger. 2 ml of the 0.5% ropivacaine slowly injected after negative aspiration of blood was confirmed. Inserting the needle 1 cm above the inner canthus, targeting the junction of the orbit and the nasal bone, performed infratrochlear nerve block. After negative aspiration of blood, 1 ml of the 0.5% ropivacaine was injected. Contralateral nerve block was performed in the same manner.
  Arms: Nerve Block Group
Other: without any nerve block — Patients receiving general anesthesia without Infraorbital and Infratrochlear nerve block.
  Other Names: nerve block with 0.5% ropivacaine
  Arms: Control Group

SUMMARY:
The endoscopic binostril transnasal transsphenoidal resection of pituitary procedures often cause intense pain which is difficult to suppress at the depth of conventional general anesthesia, resulting in severe hemodynamic fluctuations in patients. Infraorbital and infratrochlear nerve block can block the pain signal caused by the endoscopic binostril transnasal transsphenoidal resection of pituitary theoretically, which has been proven to provide satisfactory analgesia after septorhinoplasty. However, whether bilateral infraorbital and infratrochlear nerve block can provide stable hemodynamics and reduce the hemodynamic fluctuation the patients undergoing endoscopic binostril transnasal transsphenoidal resection of pituitary remains unclear.

DETAILED DESCRIPTION:
Surgical stimulation is one of the important factors leading to hemodynamic fluctuation and affecting postoperative recovery quality. The endoscopic binostril transnasal transsphenoidal resection of pituitary procedures often cause intense pain because of there were numerous nerve endings at the surgical site which is originated from branches of the trigeminal nerve (including infraorbital and infratrochlear nerve). It's difficult to suppress intraoperative stimulation at the depth of conventional general anesthesia, resulting in severe hemodynamic fluctuations in patients. It's reported that pterygomaxillary fossa block can inhibit hypertension caused by surgical procedures, however the block may cause complications because of its complicated operations. Infraorbital and infratrochlear nerve block can block the pain signal caused by the endoscopic binostril transnasal transsphenoidal resection of pituitary theoretically, which has been proven to provide satisfactory analgesia after septorhinoplasty. However, whether bilateral infraorbital and infratrochlear nerve block can reduce the pain in the patients undergoing endoscopic binostril transnasal transsphenoidal resection of pituitary remains unclear. Therefore, the investigators propose the hypothesis that preoperative bilateral infraorbital and infratrochlear nerve block could effectively reduce the pain in patients undergoing endoscopic binostril transnasal transsphenoidal resection of pituitary. The objective of this study is to observe the heart rate and blood pressure at a specific point in time during the operation and pain at 2, 8, 24, 48 hours postoperatively between adult patients receiving or not receiving bilateral infraorbital and infratrochlear nerve block.

ELIGIBILITY:
Inclusion Criteria:

* 1. Elective endoscopic binostril transnasal transsphenoidal resection
* 2. Patients aged between 18 and 65.
* 3. American Society of Anesthesiologists (ASA) physical status I, Ⅱ and III

Exclusion Criteria:

* 1. Emergency operation.
* 2. Patients allergic to ropivacaine.
* 3. Infection nearby the puncture point.
* 4. Patients with preoperative usage of sedative and analgesic drugs with history of alcohol abuse.
* 5. Patient with renal insufficiency or hepatic failure.
* 6. Patients who have undergone craniotomy in the recent 6 months.
* 7. Pregnant or lactating women, being participating in other studies.
* 8. Patients unable to cooperate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-28 (Estimated); Study Completion 2023-09-28 (Estimated)

PRIMARY OUTCOMES:
mean arterial pressure (MAP) before nerve block | before nerve block
  mean arterial pressure (MAP) before nerve block
heat rate (HR) before nerve block | before nerve block
  heat rate (HR) before nerve block
MAP within 10 minutes after nerve block | within 10 minutes after nerve block
  MAP within 10 minutes after nerve block
HR within 10 minutes after nerve block | within 10 minutes after nerve block
  HR within 10 minutes after nerve block
MAP before nasal mucosal dissection | before nasal mucosal dissection
  MAP before nasal mucosal dissection
HR before nasal mucosal dissection | before nasal mucosal dissection
  HR before nasal mucosal dissection
MAP immediately after nasal mucosal dissection | immediately after nasal mucosal dissection
  MAP immediately after nasal mucosal dissection
HR immediately after nasal mucosal dissection | immediately after nasal mucosal dissection
  HR immediately after nasal mucosal dissection
MAP before septum resection | before septum resection
  MAP before septum resection
HR before septum resection | before septum resection
  HR before septum resection
MAP immediately after septum resection | immediately after septum resection
  MAP immediately after septum resection
HR immediately after septum resection | immediately after septum resection
  HR immediately after septum resection
MAP before sella bone resection | before sella bone resection
  MAP before sella bone resection
HR before sella bone resection | before sella bone resection
  HR before sella bone resection
MAP after sella bone resection | before sella bone resection
  MAP after sella bone resection
HR immediately after sella bone resection | immediately after sella bone resection
  HR immediately after sella bone resection
MAP before dural incision of sella | before dural incision of sella
  MAP before dural incision of sella
HR before dural incision of sella | before dural incision of sella
  HR before dural incision of sella
MAP immediately after dural incision of sella | immediately after dural incision of sella
  MAP immediately after dural incision of sella
HR immediately after dural incision of sella | immediately after dural incision of sella
  HR immediately after dural incision of sella
MAP before exploration of pituitary fossa | before exploration of pituitary fossa
  MAP before exploration of pituitary fossa
HR before exploration of pituitary fossa | before exploration of pituitary fossa
  HR before exploration of pituitary fossa
MAP immediately after exploration of pituitary fossa | immediately after exploration of pituitary fossa
  MAP immediately after exploration of pituitary fossa
HR immediately after exploration of pituitary fossa | immediately after exploration of pituitary fossa
  HR immediately after exploration of pituitary fossa

SECONDARY OUTCOMES:
numerical rating scale (NRS) score when patient enters post-anaesthesia care unit (PACU) (immediately after surgery) | when patient enters PACU (immediately after surgery)
  numerical rating scale (NRS) score when patient enters PACU (immediately after surgery). The participants subjectively determine the patient's pain scores using a 0 to 10 NRS (0 = no pain; 10 = unbearable pain), to evaluate the efficacy of the modified method.
numerical rating scale (NRS) score before patient leaves PACU | before patient leaves PACU
  numerical rating scale (NRS) score before patient leaves PACU. The participants subjectively determine the patient's pain scores using a 0 to 10 NRS (0 = no pain; 10 = unbearable pain), to evaluate the efficacy of the modified method.
NRS 2 hours after surgery | 2 hours after surgery
  NRS 2 hours after surgery. The participants subjectively determine the patient's pain scores using a 0 to 10 NRS (0 = no pain; 10 = unbearable pain), to evaluate the efficacy of the modified method.
NRS 8 hours after surgery | 8 hours after surgery
  NRS 8 hours after surgery. The participants subjectively determine the patient's pain scores using a 0 to 10 NRS (0 = no pain; 10 = unbearable pain), to evaluate the efficacy of the modified method.
NRS 24 hours after surgery | 24 hours after surgery
  NRS 24 hours after surgery. The participants subjectively determine the patient's pain scores using a 0 to 10 NRS (0 = no pain; 10 = unbearable pain), to evaluate the efficacy of the modified method.
NRS 48 hours after surgery | 48 hours after surgery
  NRS 48 hours after surgery. The participants subjectively determine the patient's pain scores using a 0 to 10 NRS (0 = no pain; 10 = unbearable pain), to evaluate the efficacy of the modified method.
quality of recovery Scale: Quality of Recovery-15 (QoR-15) 1 day after surgery | 1 day after surgery
  quality of recovery Scale (QoR-15): QoR-15 1 day after surgery. QoR-15 contains the five aspects (physiological comfort, physiological independence, psychological support, emotion and pain), which can evaluate postoperative recovery quality.
quality of recovery Scale: QoR-15 3 days after surgery | 3 days after surgery
  quality of recovery Scale: QoR-15 3 days after surgery. QoR-15 contains the five aspects (physiological comfort, physiological independence, psychological support, emotion and pain), which can evaluate postoperative recovery quality.
quality of recovery Scale: QoR-15 7 days after surgery | 7 days after surgery
  quality of recovery Scale: QoR-15 7 days after surgery. QoR-15 contains the five aspects (physiological comfort, physiological independence, psychological support, emotion and pain), which can evaluate postoperative recovery quality.

OTHER OUTCOMES:
incidence of postoperative nausea and vomiting (PONV) within 24 hours | within 24h after surgery
  within 24 hours after surgery, the investigators record the number of patients who suffer from PONV, and then calculate the incidence as: the number of patient suffering from PONV/the total number in corresponding group
incidence of postoperative nausea and vomiting (PONV) within 48 hours | within 48 hours after surgery
  within 48 hours after surgery, the investigators record the number of patients who suffer from PONV, and then calculate the incidence as: the number of patient suffering from PONV/the total number in corresponding group
Ramsay sedation scale (RSS) when patient enters PACU (immediately after surgery) | when patient enters PACU (immediately after surgery)
  Ramsay sedation scale (RSS) when patient enters PACU (immediately after surgery). The participants subjectively determine the patient's sedation scores using a 1 to 6 RSS (1=fidgety, 2-4=sedation satisfaction, 5-6=excessive sedation).
Ramsay sedation scale (RSS) before patient leaves PACU | before patient leaves PACU
  Ramsay sedation scale (RSS) before patient leaves PACU. The participants subjectively determine the patient's sedation scores using a 1 to 6 RSS (1=fidgety, 2-4=sedation satisfaction, 5-6=excessive sedation).
Ramsay sedation scale (RSS) 2 hours after surgery | 2 hours after surgery
  Ramsay sedation scale (RSS) 2 hours after surgery. The participants subjectively determine the patient's sedation scores using a 1 to 6 RSS (1=fidgety, 2-4=sedation satisfaction, 5-6=excessive sedation).
Ramsay sedation scale (RSS) 8 hours after surgery | 8 hours after surgery
  Ramsay sedation scale (RSS) 8 hours after surgery. The participants subjectively determine the patient's sedation scores using a 1 to 6 RSS (1=fidgety, 2-4=sedation satisfaction, 5-6=excessive sedation).
Ramsay sedation scale (RSS) 24 hours after surgery | 24 hours after surgery
  Ramsay sedation scale (RSS) 24 hours after surgery. The participants subjectively determine the patient's sedation scores using a 1 to 6 RSS (1=fidgety, 2-4=sedation satisfaction, 5-6=excessive sedation).
Ramsay sedation scale (RSS) 48 hours after surgery | 48 hours after surgery
  Ramsay sedation scale (RSS) 48 hours after surgery. The participants subjectively determine the patient's sedation scores using a 1 to 6 RSS (1=fidgety, 2-4=sedation satisfaction, 5-6=excessive sedation).
operation time | from the time of surgery beginning until end time of surgery
  from the time of surgery beginning until end time of surgery
anesthesia time | from the time of anesthesia beginning until end time of anesthesia
  from the time of anesthesia beginning until end time of anesthesia
awakening time | from the time of anesthesia end until the time of patient awaken
  from the time of anesthesia end until the time of patient awaken
PACU staying time | from the time of patient coming in PACU until the time of patient coming out PACU
  time from the time of patient coming in PACU until the time of patient coming out PACU
anesthetic dosage | during surgery
  use dosage of anesthetic drug during operation
urine volume | during surgery
  urine volume during surgery
bleeding volume | during surgery
  bleeding volume during surgery
maintenance infusion rate of remifentanil | during surgery
  infusion rate of remifentanil for maintaining effective analgesic effect during surgery
the dosage of remedial painkillers (remifentanil) | during surgery
  the dosage of remedial painkillers (remifentanil) during surgery
the dosage of remedial perdipine | during surgery
  the dosage of remedial perdipine during surgery
the dosage of remedial esmolol | during surgery
  the dosage of remedial esmolol during surgery
the time of initial administration of remedial antiemetics within 48 hours | within 48 hours after surgery
  the time of initial administration of remedial antiemetics within 48 hours after surgery
the dosage of remedial antiemetics within 48 hours | within 48 hours after surgery
  the dosage of remedial antiemetics within 48 hours after surgery
incidence of hematoma at the block point in both two groups within 24 hours | within 24 hours after surgery
  within 24 hours after operation, the investigators record the number of patients who suffer from hematoma at the block point, and then calculate the incidence as: the number of patient suffering from hematoma at the block point/the total number in corresponding group
incidence of infection at the block point in both two groups within 24 hours | within 24 hours after surgery
  within 24 hours after operation, the investigators record the number of patients who suffer from infection at the block point, and then calculate the incidence as: the number of patient suffering from infection at the block point/the total number in corresponding group
incidence of local anesthetic toxicity in both two groups within 24 hours | within 24 hours after surgery
  within 24 hours after operation, the investigators record the number of patients who suffer from local anesthetic toxicity, and then calculate the incidence as: the number of patient suffering from local anesthetic toxicity/the total number in corresponding group

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China